CLINICAL TRIAL: NCT00142610
Title: Effect of Alpha Tocopherol and Ascorbate Supplementation on Airway Antioxidant Levels in Allergic Asthmatics
Brief Title: The Role of Vitamins E and C in Maintaining Lung Health in People With Asthma
Acronym: VITAS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, David B. Peden, MD, Director Enviro Med Asthma & Lung Biology, University of North Carolina, Chapel Hill
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P01AT002620-02 (NIH); P01AT002620-02 (NIH); Project #1; Grant ID - PO1-AT002620-02
Record Dates: First submitted 2005-09-01; First posted 2005-09-02 (Estimated); Last update posted 2013-03-04 (Estimated); Status verified 2013-02

CONDITIONS: Asthma
Keywords: alpha tocopherol; vitamin E; ascorbate; vitamin C; antioxidant; allergic; asthma
MeSH Terms: conditions — Asthma | interventions — Vitamins; Ascorbic Acid; Vitamin E

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- vitamin (Experimental): 500 mg alpha tocopherol combined with 2,000 mg of ascorbate, each orally administered daily for 12 weeks
  Interventions: Dietary Supplement: Vitamin
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Vitamin

INTERVENTIONS:
Dietary Supplement: Vitamin — This is designed as a placebo controlled study of 500 mg alpha tocopherol combined with 2,000 mg of ascorbate, each orally administered daily for 12 weeks, on airway antioxidant levels in asthmatics.
  Other Names: Vitamin C; Vitamin E

SUMMARY:
This study will determine if airway antioxidant levels in allergic asthmatics are enhanced with a combination of vitamin E and vitamin C therapy.

DETAILED DESCRIPTION:
Eosinophils and neutrophils are inflammatory cells located in the airways and lungs. When they are activated, they generate oxidants, which irritates the mucosal cells in the airways. As a result, mucus develops in the lungs. Allergens can activate the inflammatory cells, thereby worsening the symptoms of asthma in allergic asthmatics. Vitamins E (alpha-tocopherol) and C (ascorbate) have been shown to decrease asthma exacerbation associated with exposure to ozone. Enhancing antioxidant and anti-inflammatory defenses in the airways and lungs is a promising approach for treating respiratory diseases aggravated by allergies. This study will determine if airway antioxidants in allergic asthmatics are enhanced with a combination of vitamin E and vitamin C therapy.

Participants in this double-blind study will be randomly assigned to receive either a combination of alpha-tocopherol and ascorbate or placebo. Treatments will be administered daily for 12 weeks. Baseline assessments will measure airway and circulating antioxidant levels, inflammatory cells, lung function, respiratory symptoms, and methacholine reactivity. Allergy skin tests will also be performed to determine the state of atopy, which is a hereditary predisposition toward developing certain hypersensitivity reactions. Following baseline assessments, lung assessments will be conducted weekly for 12 weeks, sputum and blood samples will be collected bi-weekly, and methacholine reactivity will be assessed at Weeks 6 and 12.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed allergy to at least one of the following allergen preparations: house dust mite f; house dust mite p; cockroach; tree mix; grass mix; weed mix; mold mix 1; mold mix 2; rat; mouse; guinea pig; rabbit; cat; or dog
* Oxygen saturation greater than 94% at baseline
* Systolic blood pressure between 150 and 90 mm Hg, diastolic blood pressure between 90 and 60 mm Hg
* Physician-diagnosed asthma or history of episodic wheezing, chest tightness, or shortness of breath consistent with asthma
* Airway reactivity as determined by either a provocative concentration of methacholine producing a 20% fall in FEV1 (PC20 methacholine) of less than 10 mg/ml by the method used or 12% reversibility of baseline lung function with albuterol therapy for two of the three measures: FVC, FEV1, and FEF25-75%
* Agree to discontinue use of vitamin supplements for the duration of the study
* On a stable regimen of maintenance asthma therapy that has not changed within the month prior to participation

Exclusion Criteria:

* Chronic medical condition that may make vitamin E and vitamin C treatment medically inadvisable (e.g., significant cardiovascular disease, diabetes requiring medication, chronic kidney disease, chronic thyroid disease, or coagulation defects)
* History of kidney stones
* Use of anticoagulants (e.g., warfarin, heparin, or clopindogrel)
* Pregnant or breastfeeding
* Use of inhaled steroids, cromolyn, or leukotriene inhibitors (Montelukast or Zafirkulast) for at least one month is not criteria for exclusion.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2005-08; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Sputum cell ascorbate and alpha-tocopherol levels; measured bi-weekly and at Week 12 | measurements have been made alalysis still occuring

SECONDARY OUTCOMES:
Methacholine reactivity; measured at Weeks 6 and 12 | measure finished, analysis continues
Lung function and symptom scores; measured weekly and at Week 12 | measuremet finished, analysis continues

CONTACTS AND LOCATIONS:
Overall Officials: David B. Peden, MD, MS, Principal Investigator — Center for Environmental Medicine, Asthma, and Lung Biology
Locations (1):
- UNC EPA, Chapel Hill, North Carolina, United States

REFERENCES:
- See also: Center for Environmental Medicine, Asthma, and Lung Biology — http://www.med.unc.edu/cemalb